CLINICAL TRIAL: NCT03511222
Title: A Phase IB Trial of Vorolanib (X-82) Combined With Checkpoint Inhibitors in Patients With Solid Tumors
Brief Title: Vorolanib (X-82) Combined With Checkpoint Inhibitors in Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Collaborators: Xcovery Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201806087
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Solid Tumor; Hepatocellular Carcinoma; Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Stomach Neoplasms | interventions — vorolanib; Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Dose Escalation: Vorolanib + Nivolumab (Experimental): * Vorolanib is an oral drug which will be administered daily on an outpatient basis at the assigned dose level.
  * Patients receiving nivolumab will get it on an outpatient basis as a 30-minute intravenous infusion at a dose of 480 mg on Day 1 of each 28-day cycle
  * In light of immunotherapy approach, treatment beyond progression is allowed as long as patient has clinical stability. Patients can stay on the regimen unless excessive toxicity or clinical or radiographic disease progression per RECIST
  Interventions: Drug: Vorolanib; Drug: Nivolumab
- Dose Escalation: Vorolanib + Pembrolizumab (Experimental): * Vorolanib is an oral drug which will be administered daily on an outpatient basis at the assigned dose level
  * Patients receiving pembrolizumab will get it on an outpatient basis as a 30-minute (-5/+10 minutes) intravenous infusion at a dose of 200 mg on Day 1 of each 21-day cycle
  * In light of immunotherapy approach, treatment beyond progression is allowed as long as patient has clinical stability. Patients can stay on the regimen unless excessive toxicity or clinical or radiographic disease progression per RECIST
  Interventions: Drug: Vorolanib; Drug: Pembrolizumab
- Vorolanib + Nivolumab (Small Cell Lung Cancer) (Experimental): * Vorolanib is an oral drug which will be administered daily on an outpatient basis at 300 mg daily
  * Patients receiving nivolumab will get it on an outpatient basis as a 30-minute intravenous infusion at a dose of 480 mg on Day 1 of each 28-day cycle
  * In light of immunotherapy approach, treatment beyond progression is allowed as long as patient has clinical stability. Patients can stay on the regimen unless excessive toxicity or clinical or radiographic disease progression per RECIST
  Interventions: Drug: Vorolanib; Drug: Nivolumab

INTERVENTIONS:
Drug: Vorolanib — Patients should take vorolanib at approximately the same time every day with food.
  Other Names: X-82
Drug: Nivolumab — Standard of care
  Other Names: Opdivo
  Arms: Dose Escalation: Vorolanib + Nivolumab; Vorolanib + Nivolumab (Small Cell Lung Cancer)
Drug: Pembrolizumab — Standard of care
  Other Names: Keytruda
  Arms: Dose Escalation: Vorolanib + Pembrolizumab

SUMMARY:
The investigators hypothesize that vorolanib in combination with checkpoint inhibitors (pembrolizumab for gastric/gastroesophageal (GE) junction cancers and nivolumab for hepatocellular carcinoma (HCC)) may improve immunotherapy efficacy by overcoming treatment resistance of checkpoint inhibitors in gastrointestinal (GI) cancers.

ELIGIBILITY:
Inclusion Criteria:

* Dose escalation cohort: histologically or cytologically confirmed diagnosis of a solid tumor that can be treated with either pembrolizumab or nivolumab as part of standard of care or whom no standard of therapy exists except pembrolizumab or nivolumab
* SCLC cohort: histologically or cytologically confirmed diagnosis of small cell lung cancer whose disease progressed on platinum-based chemotherapy or refused chemotherapy
* Evidence of measurable disease per RECIST 1.1. Measurable disease is defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 2,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN (≤ 5 x IULN for patients with liver metastases or hepatocellular carcinoma (HCC))
  * Creatinine ≤ 1.5 x IULN OR measured or calculated creatinine clearance ≥ 50 mL/min for patients with creatinine levels > 1.5 x IULN
  * Urine protein ≤1+ or urine protein to creatinine ratio ≤ 1; if UPC ratio is >1 on urinalysis, then 24-hour urine collection from protein must be obtained and level must be <1,000 mg for patient enrollment.
  * aPTT and either INR or PT ≤ 1.5 x ILUN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* Patients receiving therapeutic non-Coumadin anticoagulation are eligible, provided they are on a stable dose (per investigator judgment) of anticoagulant.
* Patients with treated/stable brain metastases, defined as patients who have received prior therapy for their brain metastases and whose CNS disease is radiographically stable at study entry, are eligible. Patients with clinically evident CNS hemorrhage on scans are excluded.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 31 weeks after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Presence of a concurrent active, incurable malignancy that may alter the outcome of the treatment for disease under treatment as determined by the treating physician.
* Receiving any other investigational agents within 21 days or 5 half-lives (whichever is shorter) prior to the first dose of study drug.
* Prior PD-1 or PD-L1 inhibitor therapy, or prior therapy with anti-PD-L2 or anti-CTLA-4 inhibitor, or any other drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to vorolanib, nivolumab or pembrolizumab (as applicable), any monoclonal antibody, or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection.
* Has a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses ≤ 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). A brief course of corticosteroids for prophylaxis (e.g. contrast dye allergy) or for treatment of non-autoimmune conditions (e.g. delayed-type hypersensitivity reaction caused by contact allergens) is permitted.
* Toxicities from prior therapy must have resolved to G1 or less prior to the first dose of study drug except those deemed not clinically significant per PI.
* Active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids. This includes but is not limited to: history of immune-related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as SLE, connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome. Patients with vitiligo or endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome, and psoriasis controlled with topical medication, and patients with positive serology, such as antinuclear antibodies (ANA) or anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible. Patients with type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, or conditions not expected to recur in the absence of an external trigger (precipitating event) are eligible.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* History of clinically significant bleeding.
* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, GI obstruction, and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study.
* Inability to swallow or retain oral medications or the presence of active GI disease or other conditions that will interfere significantly with the absorption, distribution, metabolism, or excretion of vorolanib.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 24 hours of study entry.
* Active hepatitis B or hepatitis C. Note: no testing for hepatitis B or C is required unless mandated by local health authority.
* Has a known history of active tuberculosis.
* Known HIV-positivity.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist) are live attenuated vaccines and are not allowed.
* Major surgery within the last 4 weeks; minor surgery within the last 2 weeks.
* Any radiotherapy within 3 weeks except palliative stereotactic body radiation therapy (SBRT) within 2 weeks.
* Prior anti-cancer therapy given within 21 days or 5 half-lives (whichever is shorter)
* Chemotherapy given on the weekly basis with limited potential for delayed toxicity within the last 2 weeks.
* Concurrent use of any medications or substances (e.g. herbal supplement or food) known to be a strong inhibitor or strong inducer of CYP3A4.
* Symptomatic arterial peripheral vascular disease or significant cardiovascular disease or condition including:

  * Congestive heart failure (CHF) currently requiring therapy.
  * Class III or IV cardiovascular disease according to the New York Heart Association (NYHA) Functional Criteria.
  * Need for antiarrhythmic medical therapy for a ventricular arrhythmia.
  * Severe conduction disturbance (e.g. 3rd degree heart block).
  * Unstable angina pectoris (i.e. last episode ≤ 6 months prior to first dose of protocol-indicated treatment).
  * Uncontrolled (per investigator judgment) hypertension.
  * Myocardial infarction within 6 months prior to starting trial treatment.
  * QTcF >450 ms in men, or >470 ms in women.
* Deep vein thrombosis or pulmonary embolism ≤ 4 weeks before first dose of protocol-indicated treatment, unless adequately treated and stable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) of vorolanib plus pembrolizumab | Completion of enrollment to Dose Escalation cohorts (estimated to be 13 months)
  -The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity during the first cycle. Dose escalations will proceed for both nivolumab and pembrolizumab until the MTD or highest dose level (level 2), which is defined as RP2D.
Recommended phase II dose (RP2D) of vorolanib plus nivolumab | Completion of enrollment to Dose Escalation cohorts (estimated to be 13 months)
  -The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity during the first cycle. Dose escalations will proceed for both nivolumab and pembrolizumab until the MTD or highest dose level (level 2), which is defined as RP2D.

SECONDARY OUTCOMES:
Safety and toxicity of vorolanib plus pembrolizumab as measured by the number and type of adverse events experienced by participant | 30 days after completion of treatment (estimated to be 7 months)
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.
Safety and toxicity of vorolanib plus nivolumab as measured by the number and type of adverse events experienced by participant | 30 days after completion of treatment (estimated to be 7 months)
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Nusayba A Bagegni, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bagegni NA, Park H, Kraft K, O-Toole M, Gao F, Waqar SN, Ratner L, Morgensztern D, Devarakonda S, Amin M, Baggstrom MQ, Liang C, Selvaggi G, Wang-Gillam A. Phase 1b trial of anti-VEGF/PDGFR vorolanib combined with immune checkpoint inhibitors in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2022 Apr;89(4):487-497. doi: 10.1007/s00280-022-04406-6. Epub 2022 Mar 5. PMID 35247086
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu